CLINICAL TRIAL: NCT02695238
Title: Trial of Prophylactic Manual Rotation of Persistent Occiput Posterior Presentation During the Early Second Stage of Labor to Reduce Operative Delivery: a Prospective Multicenter Randomized Control Trial
Acronym: PROPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00225-44
Record Dates: First submitted 2016-01-29; First posted 2016-03-01 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Persistent Occipital Posterior Presentation During Labor Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prophylactic manual rotation group (Experimental): During persistent occipital posterior presentation during the second stage of labor, prophylactic manual rotation will be performed.
  Interventions: Procedure: Prophylactic Manual Rotation of persistent occipital posterior presentation
- No prophylactic manual rotation group (No Intervention): During persistent occipital posterior presentation during the second stage of labor, expectant management for delevery will be performed

INTERVENTIONS:
Procedure: Prophylactic Manual Rotation of persistent occipital posterior presentation — prophylactic manual rotation of persistent occipital posterior presentation on operative delivery will be performed in the experimental group
  Arms: prophylactic manual rotation group

SUMMARY:
Superiority multicenter prospective randomized study on operative delivery (instrumental delivery or caesarean section) of prophylactic manual rotation in case of persistent occipital posterior presentation during the second stage of labor compared to expectant management. A 15% reduction of operative delivery (instrumental delivery or caesarean section) is attempt in the prophylactic manual rotation group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Singleton pregnancy
* Term ≥ 37 weeks of gestation
* Early second stage of labor
* Rupture membranes
* Persistent occiput posterior position confirmed by ultrasound
* Epidural anesthesia
* Patient who agree to participate and sign consent form

Exclusion Criteria:

* Age < 18 years
* Term < 37 weeks of gestation
* Vaginal and instrumental Delivery maternal contraindication
* Antecedent of perineal injury type IV
* Sensitive perineum
* Crohn's disease with vaginal delivery contraindication
* Instrumental fetal contraindication
* Non reassuring fetal heart with impossibility of optimal maternal information
* Known fetal malformation
* Previous ceaserean section
* Non cephalic presentation
* Not affiliated to social security

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who will have a caesarean section or an instrumental delivery in each groups. | 4 hours

SECONDARY OUTCOMES:
Number of patients with episiotomy, perineal lacerations from the 1st to the 4rth degree anglo-saxon classification | 4 hours
Number of patients who will have bladder, urinary or bowel injuries during caesarean section | 5 hours maximum
Number of patients with post-partum hemorrhage defined by blood loss more than 500mL | 5 hours maximum

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Blanc J, Castel P, Mauviel F, Baumstarck K, Bretelle F, D'Ercole C, Haumonte JB. Prophylactic manual rotation of occiput posterior and transverse positions to decrease operative delivery: the PROPOP randomized clinical trial. Am J Obstet Gynecol. 2021 Oct;225(4):444.e1-444.e8. doi: 10.1016/j.ajog.2021.05.020. Epub 2021 May 24. PMID 34033811